CLINICAL TRIAL: NCT00169403
Title: Pallidal Stimulation in Patients With Idiopathic Generalised Dystonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: University Hospital, Tours (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P000201
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2005-09

CONDITIONS: Dystonia
Keywords: Idiopathic dystonia; deep brain stimulation; globus pallidus; generalised Idiopathic dystonia
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation

SUMMARY:
Pallidal stimulation is effective in patients with generalised idiopathic dystonia. The aim of this study is to:

1. evaluate the efficacy and safety of this treatment in patients with idiopathic generalised dystonia, 3 years after surgery and
2. assess the recurrence of the motor symptoms after the switch off.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic generalised dystonia
* Pallidal stimulation

Exclusion Criteria:

* Mini-mental status (MMS) < 24
* Severe psychiatric disorder

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marie Vidailhet, MD, PhD, Study Director — Hôpital Saint-Antoine
Locations (1):
- Centre d'Investigation Clinique-Hôpital Pitié-Salpetriere, Paris, France

REFERENCES:
- [Result] Vidailhet M, Vercueil L, Houeto JL, Krystkowiak P, Benabid AL, Cornu P, Lagrange C, Tezenas du Montcel S, Dormont D, Grand S, Blond S, Detante O, Pillon B, Ardouin C, Agid Y, Destee A, Pollak P; French Stimulation du Pallidum Interne dans la Dystonie (SPIDY) Study Group. Bilateral deep-brain stimulation of the globus pallidus in primary generalized dystonia. N Engl J Med. 2005 Feb 3;352(5):459-67. doi: 10.1056/NEJMoa042187. PMID 15689584